CLINICAL TRIAL: NCT01132521
Title: Multicenter, Double-bind, Randomised, Placebo Controlled Study of Ulinastatin in Severe Acute Pancreatitis
Brief Title: Ulinastatin in Severe Acute Pancreatitis
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Revised project
Sponsor: Techpool Bio-Pharma Co., Ltd. (Industry)
Collaborators: Peking Union Medical College Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The first clinical college of harbin medical university (Unknown); The First Affiliated Hospital with Nanjing Medical University (Other); West China Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UTI/SAP-S
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Pancreatitis
Keywords: ulinastatin; severe acute pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — urinastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ulinastatin group (Experimental): Regular treatments plus ulinastatin. Resolved 4 vials of drugs in 100ml physiological saline solution, intravenously infused for 1-2h, tid, for continuous 7 days.
  Interventions: Drug: ulinastatin
- placebo group (Placebo Comparator): Regular treatment plus placebo. Resolved 4 vials of drugs in 100ml physiological saline solution, intravenously infused for 1-2h, tid, for continuous 7 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ulinastatin — Resolved 4 vials of drugs in 100ml physiological saline solution, intravenously infused for 1-2h, tid, for continuous 7 days.
  Other Names: UTI; urinary trypsin inhibitor; bikunin
  Arms: ulinastatin group
Drug: placebo — Resolved 4 vials of drugs in 100ml physiological saline solution, intravenously infused for 1-2h, tid, for continuous 7 days.
  Arms: placebo group

SUMMARY:
This study aims to evaluate the effect of ulinastatin in the treatment and prevention of organ failure in severe acute pancreatitis.

DETAILED DESCRIPTION:
About 20% of patients with acute pancreatitis have a severe course, and 10-15% of those with severe acute pancreatitis (SAP) die. Despite improvements in intensive care treatment during past few decades, effective therapies for acute pancreatitis are still limited.

Early deaths (within the first week) due to severe acute pancreatitis are generally caused by massive inflammatory responses which result in multiple organ failure. Although the exact mechanisms which trigger the inflammatory processes are not completely understood, it is generally accepted that autodigestion and activated leukocytes play important roles in the pathogenesis of acute pancreatitis. Activation of digestive enzymes causes pancreatic injury and results in an inflammatory response that is out of proportion to the response of other organs to a similar insult. The acute inflammatory response itself causes substantial tissue damage and may progress beyond the pancreas to a systemic inflammatory response syndrome, multi organ failure, or death.

UTI is a multivalent Kunitz-type serine protease inhibitor that is found in human urine and blood, it can stabilize lysosome membrane and inhibit lysosome function, inhibit the various enzymes and inflammatory response. Previous study proved that it protects against SIRS pathophysiology and subsequent organ damage induced via the modulation of the proinflammatory mediator, as well as chemokines. UTI has been widely used for the treatment and prevention of multiple organ failure in China, but there is few randomized, placebo controlled trial on ulinastatin. A large multicenter, randomized study is warranted. In this study, we aim to evaluate the effect of ulinastatin in the treatment and prevention of organ failure in severe acute pancreatitis with regular treatment in an add-on trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe acute pancreatitis , severe acute pancreatitis adapted from the Atlanta classification:

Early Prognostic Signs: Ramson signs ≥3, APACHE II score ≥8 Organ Failure and/or Local Complications: Necrosis, Abscess, Pseudocyst;

* Admission within 72h after onset of symptoms of pancreatitis
* 18-70 years old
* Signed the informed consent form

Exclusion Criteria:

* Pre-existing chronic renal insufficiency requiring hemodialysis or peritoneal dialysis
* pre existing heart dysfunction or NYHA classification score above III
* pregnancy or lactation
* Allergy for ulinastatin
* Received an investigational drug or device within 90 days prior to entering study
* serious mentally-ill patients including dementia
* On the verge of death (estimated to be mortal in 12h).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
multiple organ dysfunction score | 8 days
onset of (multiple) organ failure after randomized | 8 days

SECONDARY OUTCOMES:
mortality | 8 days, 14 days and 28 days
Incidence of complications | 8 days, 14 days and 28 days
APACHE Ⅱ score | 8 days
Need for surgical intervention | From admission to discharge
Hospital stay and ICU stay | From admission to discharge
CT-scan score | 8 days, 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Yupei Zhao, MD, Study Chair — Peking Union Medical College Hospital; Chunyou Wang, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (6):
- China (6):
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Clinical College of Harbin University, Harbin, Heilongjiang
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - West China Hospital, Chengdu, Sichuan
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wang CY, Zhao YP. Progress of therapeutic effect in severe acute pancreatitis: Mini-review of treatment viewpoints and technique improvements. Chin J Surg 44(13): 872-4, 2006. (Article in Chinese)
- [Result] Maehara K, Kanayama N, Halim A, el Maradny E, Oda T, Fujita M, Terao T. Down-regulation of interleukin-8 gene expression in HL60 cell line by human Kunitz-type trypsin inhibitor. Biochem Biophys Res Commun. 1995 Jan 26;206(3):927-34. doi: 10.1006/bbrc.1995.1131. PMID 7832806
- [Result] Tsujino T, Komatsu Y, Isayama H, Hirano K, Sasahira N, Yamamoto N, Toda N, Ito Y, Nakai Y, Tada M, Matsumura M, Yoshida H, Kawabe T, Shiratori Y, Omata M. Ulinastatin for pancreatitis after endoscopic retrograde cholangiopancreatography: a randomized, controlled trial. Clin Gastroenterol Hepatol. 2005 Apr;3(4):376-83. doi: 10.1016/s1542-3565(04)00671-8. PMID 15822043
- See also: Related Info — http://pir.georgetown.edu/cgi-bin/ipcSF?id=PIRSF001622